CLINICAL TRIAL: NCT06853938
Title: Optimizing Transhumeral Osseointegration Prosthesis Control
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00140248
Record Dates: First submitted 2025-02-24; First posted 2025-03-03 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Transhumeral Amputation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Persons with transhumeral amputation who receive an enhanced muscle training protocol and fitting with a myoelectric (muscle signal-controlled) device after receiving osseointegrated implant and targeted muscle reinnervation.
  Interventions: Device: Myoelectric prosthesis

INTERVENTIONS:
Device: Myoelectric prosthesis — The interventions in this study are (1) an enhanced muscle training protocol and (2) fitting with a myoelectric (muscle signal-controlled) prosthetic device after receiving an osseointegrated implant and targeted muscle reinnervation.

SUMMARY:
Upper limb amputation above the elbow results in a significant loss of function. There have been many advancements in surgery and prosthetic devices to restore arm function, but many people still reject upper limb prostheses. This is due to difficulties with how the socket fits and poor control of the device. Above-elbow prostheses are particularly challenging to use for several reasons. The socket must go all the way into the shoulder for stability. To hold the prosthesis onto the remaining arm, there needs to be a strap across the chest and shoulder. The prosthesis can be heavy, and the socket can slip or move around. This makes it hard to use muscle signals in the residual limb to control advanced prosthetic devices. People with limb loss are interested in advanced prostheses to use them reliably for day-to-day activities.

Bone-anchored prostheses (BAPs) are a new approach. They are for people with upper limb loss who can't use socket prostheses. The surgery involves putting a titanium rod into the remaining bone, which, over time, joins with the bone. This implant extends through the skin. It enables the direct attachment of the prosthetic parts (like the elbow and hand). With BAPs, there is no need for a socket. Also, there is a well-known surgery called "Targeted muscle reinnervation" (TMR). It improves the number of arm muscle control signals. These signals are used to control myoelectric prostheses. However, after both these surgeries, there is a lack of research that shows how best to train the muscle signals to use an advanced myoelectric arm and little evidence on what factors actually improve in a person's day-to-day life when using such a prosthesis.

This study aims to implement an enhanced muscle training protocol and fitting with a myoelectric (muscle signal-controlled) device after receiving OI and TMR for above-elbow amputation, and to evaluate the outcomes over time. The goal is to understand whether these advanced prostheses improve prosthesis use and function in daily life.

ELIGIBILITY:
Inclusion Criteria:

Individuals with transhumeral amputation who:

1. are between 18 and 65 years old,
2. have been scheduled to undergo osseointegration by the Alberta Limb Osseointegration Program.
3. demonstrate adequate pain-free shoulder range of motion to perform the required tasks and have potential muscle signals for myoelectric control to be able to undertake the muscle signal training
4. willing to undergo all of the study procedures and follow-up.

Exclusion Criteria:

Individuals who:

1. are unable to comply with treatment or follow-up processes,
2. are unable to understand English sufficiently to provide full informed consent.
3. have shoulder pathology on the side of the amputation (arthritis, adhesive capsulitis, chronic rotator cuff, or musculoskeletal dysfunction) that would negatively affect the ability to perform the training and functional assessments,
4. have insufficient muscle signals to operate a myoelectric prosthesis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2028-06-14 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Prosthesis-related activity | From enrollment to the end of treatment at 12 months
  The percentage reliance on the use of the prosthesis compared to the dominant arm. Prosthesis-related activity will be measured by participants wearing activity sensor bracelets (commercially available accelerometer-based sensors, i.e. Actigraph), one on each arm, for 7 days at each assessment time point. We will calculate the sum of seconds of active use for each arm to calculate the ratio of symmetry. The primary measure will be the percentage reliance on the dominant side, calculated for when the prosthesis is worn. Measures of unilateral and bilateral activities will also be computed.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Glenrose Rehabilitation Hospital, Edmonton, Alberta
  - University of Alberta, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No